CLINICAL TRIAL: NCT00857584
Title: Effectiveness of Quetiapine XR Versus Sertraline in Acute Depression as add-on Therapy to Previous Mood Stabilizer Treatment: a Pilot Study
Brief Title: Quetiapine XR Versus Sertraline in Acute Bipolar Depression as add-on Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00058
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-03

CONDITIONS: Bipolar Disorder; Bipolar Depression
Keywords: Bipolar disorder; Bipolar depression; quetiapine; sertraline
MeSH Terms: conditions — Bipolar Disorder | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine Extended Release (Experimental): Lithium or valproate at stable doses within seric therapeutic levels
  Interventions: Drug: Extended release quetiapine (quetiapine XR); Drug: adequate mood stabilizer
- Sertraline (Active Comparator): Lithium or valproate at stable doses within seric therapeutic levels
  Interventions: Drug: Sertraline; Drug: adequate mood stabilizer

INTERVENTIONS:
Drug: Extended release quetiapine (quetiapine XR) — Flexible dose from 300 to 600 mg/d (combination of tablets of 50mg, 200mg and 300mg) oral, daily, 8 weeks length.
  Quetiapine XR was initiated at 50 mg/day and titrated to 100 mg on day 2, 200 mg on day 3, 300 mg on day 4, and flexible doses of 300 to 600 mg/d from day 5 to the end of the study.
  Other Names: SEROQUEL XR®
  Arms: Quetiapine Extended Release
Drug: Sertraline — Flexible dose from 50 to 200 mg/d (combination of tablets of 50mg and 100mg) oral, daily, 8 weeks length.
  Sertraline titration: 50 mg on day 1-3, 100 mg on day 4, and flexible doses of 50 to 200 mg/d from day 5 to the end of the study.
  Other Names: Zoloft
  Arms: Sertraline
Drug: adequate mood stabilizer — An adequate mood stabilizer treatment with lithium or valproate(defined as a serum concentration of 0.5-1.2 mEq/L or 50-100 microg/ml, respectively).

SUMMARY:
Prospective, open-label, controlled (active comparator), randomized study of 8 weeks follow-up for the evaluation of the efficacy of extended release quetiapine (quetiapine XR) versus Sertraline in addition to previous mood stabilizer treatment (lithium or valproate at stable and clinically therapeutic blood levels) in the treatment of the adult bipolar depression. This multicentric study will be featured in two sites in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Adult ambulatory patients diagnosed of bipolar disorder I or II, current depressive episode (DSM-IV-TR 4ª Ed: 296.5x or 296.89 codes)
* Have been treated with only one mood stabilizer (lithium or valproate) in optimal and stable doses during at least the previous 4 weeks to randomization
* Hamilton Depression Rating Scale (HDRS-17) total score ≥ 20 and Young Mania Rating Scale (YMRS) total score ≤ 14 at the screening and randomization visits - Informed consent signed

Exclusion Criteria:

* Patients with any axis I or II Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision (DSM-IV-TR) diagnoses different from bipolar disorder I or II - Length of current depressive episode less than 2 weeks or more than 12 months
* Having been treated with more than one mood stabilizer or any mood stabilizer other than Lithium or valproate, any antidepressant, any antipsychotic or any CP450-3A inductor/inhibitor within the 7 days period prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Research Site, Vitoria-Gasteiz, Basque Country
  - Research Site, Santander, Cantabria
  - Research Site, Zamora, Castille and León
  - Research Site, Vigo, Galicia

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine Extended Release: Extended release quetiapine (quetiapine XR) - flexible dose from 300 to 600 mg/d (combination of tablets of 50mg, 200mg and 300mg) oral, daily, 8 weeks length.
- Setraline: Sertraline - flexible dose from 50 to 200 mg/d (combination of tablets of 50mg and 100mg) oral, daily, 8 weeks length.
Period: Overall Study
Arm/Group | Quetiapine Extended Release | Setraline
Started | 14 | 13
Week 1 | 14 | 13
Week 2 | 14 | 11
Week 4 | 11 | 9
Week 8 | 10 | 8
Completed | 10 | 8
Not Completed | 4 | 5
Not completed — Lack of Efficacy | 1 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine Extended Release | Setraline | Total
Number analyzed (Participants) | 14 | 13 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.5) | 43.3 (12.6) | 46.07 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 8 | 9 | 17
Montgomery Asberg Depression Rating Scale (MADRS) total score, Continuous [Mean (Standard Deviation); unit: score on a scale] — MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms)
  score on a scale | 29.5 (5.0) [26.6 to 32.4] | 28.2 (5.8) [26.7 to 31.7] | 28.9 (5.3)
Clinical Impression Global Scale - Bipolar total score (CGI-BP-M), Continuous [Mean (Standard Deviation); unit: score on a scale] — CGI-BP-M assesses severity of clinical status. It ranges from a minimum of 1 to a maximum of 7 (higher scores indicating a greater clinical severity)
  score on a scale | 5.1 (0.7) [4.7 to 5.6] | 5.3 (0.8) [4.8 to 5.9] | 5.2 (0.8) [4.7 to 5.9]
Hamilton Anxiety Rating Scale (HARS) total score, Continuous [Mean (Standard Deviation); unit: score on a scale] — HARS assesses severity of anxiety symptoms. It ranges from a minimum of 0 to a maximum of 56 (higher scores indicating a greater severity of anxiety symptoms)
  score on a scale | 22.4 (4.03) [18.5 to 26.4] | 17.6 (4.46) [13.02 to 22.2] | 20.04 (7.38) [13.02 to 26.4]

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change From Baseline to Week 2 in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms)
Time Frame: baseline, week 2
Population: Efficacy analyses of the intent-to-treat (ITT) population (those who received at least one dose of study medication and had at least one post-baseline efficacy assessment) were conducted using ANCOVA and last observation carried forward (LOCF) methodology. Safety data were analyzed for patients who received at least one dose of study medication.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 14 | 11
score on a scale | -13.1 [-18.6 to -7.6] | -6.6 [-12.6 to -0.6]

2. Secondary Outcome: The Mean Change From Baseline to Week 1 in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: baseline, week 1
Population: Efficacy analyses of the intent-to-treat (ITT) population (those who received at least one dose of the study medication and had at least one post-baseline efficacy assessment) were conducted using ANCOVA and last observation carried forward (LOCF) methodology.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 14 | 13
score on a scale | -9.5 [-13.8 to -5.1] | -8.6 [-14.5 to -2.6]

3. Secondary Outcome: The Mean Change From Baseline to Week 4 in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: baseline, week 4
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 11 | 9
score on a scale | -16.1 [-21.4 to -10.9] | -17.7 [-25.8 to -9.7]

4. Secondary Outcome: The Mean Change From Baseline to Week 8 in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: baseline. week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 10 | 8
score on a scale | -19.4 [-24.2 to -14.5] | -18.2 [-24.8 to -11.6]

5. Secondary Outcome: The Mean Change From Baseline to Week 1 in the Clinical Impression Global Scale - Bipolar (CGI-BP-M) Total Score
Description: CGI-BP-M assesses severity of clinical status. It ranges from a minimum of 1 to a maximum of 7 ( higher scores indicating a greater clinical severity)
Time Frame: baseline, week 1
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 14 | 13
score on a scale | -0.79 [-1.47 to -0.10] | -1.08 [-2.14 to -0.02]

6. Secondary Outcome: The Mean Change From Baseline to Week 2 in the Clinical Impression Global Scale - Bipolar (CGI-BP-M) Total Score
Description: as for outcome 5
Time Frame: baseline, week 2
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 14 | 11
score on a scale | -1.36 [-2.19 to -0.52] | -1.00 [-2.20 to -0.20]

7. Secondary Outcome: The Mean Change From Baseline to Week 4 in the Clinical Impression Global Scale - Bipolar (CGI-BP-M) Total Score
Description: as for outcome 5
Time Frame: baseline, week 4
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 11 | 9
score on a scale | -2.09 [-3.19 to -0.99] | -2.56 [-4.15 to -0.97]

8. Secondary Outcome: The Mean Change From Baseline to Week 8 in the Clinical Impression Global Scale - Bipolar (CGI-BP-M) Total Score
Description: CGI-BP-M assesses severity of clinical status. It ranges from a minimum of 1 to a maximum of 7 (higher scores indicating a greater clinical severity)
Time Frame: baseline, week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 10 | 8
score on a scale | -2.9 [-4.14 to -1.66] | -2.88 [-4.25 to -1.50]

9. Secondary Outcome: The Mean Change From Baseline to Week 4 in the Hamilton Anxiety Rating Scale (HARS) Total Score
Description: HARS assesses severity of anxiety symptoms. It ranges from a minimum of 0 to a maximum of 56 (higher scores indicating a greater severity of anxiety symptoms)
Time Frame: baseline, week 4
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 11 | 9
score on a scale | -13.4 [-17.6 to -9.1] | -8.9 [-14.3 to -3.4]

10. Secondary Outcome: The Mean Change From Baseline to Week 8 in the Hamilton Anxiety Rating Scale (HARS) Total Score
Description: as for outcome 9
Time Frame: baseline, week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 10 | 8
score on a scale | -13.1 [-18.01 to -8.2] | -10.6 [-15.5 to -5.7]

11. Secondary Outcome: Number of Patients Response at Week 1
Description: Number of patients responded to the treatment at week 1, where response is defined as ≥ 50% reduction in the Montgomery Asberg Depression Rating Scale (MADRS) total score from baseline to week 1.
  MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms.
Time Frame: week 1
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 14 | 13
Participants | 4 | 4

12. Secondary Outcome: Number of Patients With Response at Week 2
Description: Number of patients responded to the treatment at week 2, where response is defined as ≥ 50% reduction in the Montgomery Asberg Depression Rating Scale (MADRS) total score from baseline to week 2.
  MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms.
Time Frame: week 2
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 14 | 11
Participants | 8 | 2

13. Secondary Outcome: Number of Patients With Response at Week 4.
Description: Number of patients responded to the treatment at week 4, where response is defined as ≥ 50% reduction in the Montgomery Asberg Depression Rating Scale (MADRS) total score from baseline to week 4.
  MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms.
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 11 | 9
Participants | 8 | 6

14. Secondary Outcome: Number of Patients With Response at Week 8.
Description: Number of patients responded to the treatment at week 8, where response is defined as ≥ 50% reduction in the Montgomery Asberg Depression Rating Scale (MADRS) total score from baseline to week 8.
  MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms.
Time Frame: week 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 10 | 8
Participants | 8 | 5

15. Secondary Outcome: Number of Patients With Remission at Week 1.
Description: Number of patients who achieved remission at week 1, where remission is defined as Montgomery Asberg Depression Rating Scale (MADRS) total score ≤ 10.
  MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms.
Time Frame: week 1
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 14 | 13
Participants | 6 | 5

16. Secondary Outcome: Number of Patients With Remission at Week 2.
Description: Number of patients who achieved remission at week 2, where remission is defined as Montgomery Asberg Depression Rating Scale (MADRS) total score ≤ 10.
  MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms.
Time Frame: week 2
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 14 | 11
Participants | 6 | 5

17. Secondary Outcome: Number of Patients With Remission at Week 4.
Description: Number of patients who achieved remission at week 4, where remission is defined as Montgomery Asberg Depression Rating Scale (MADRS) total score ≤ 10.
  MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms.
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 11 | 9
Participants | 3 | 3

18. Secondary Outcome: Number of Patients With Remission at Week 8.
Description: Number of patients who achieved remission at week 8, where remission is defined as Montgomery Asberg Depression Rating Scale (MADRS) total score ≤ 10.
  MADRS assesses severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms.
Time Frame: week 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Quetiapine Extended Release | Setraline
Number analyzed (Participants) | 10 | 8
Participants | 3 | 4

ADVERSE EVENTS:
Arm/Group | Quetiapine Extended Release | Setraline
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 12/14 | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine Extended Release (N=14) | Setraline (N=13)
Dry mouth (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0
Somnolence (Nervous system disorders) | 5 | 1
Tremor (Nervous system disorders) | 2 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Decreased libido (Psychiatric disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No